CLINICAL TRIAL: NCT03170336
Title: The Effect and Safety of Amiloride in Decreasing Proteinuria for Patients With Chronic Kidney Disease in a Prospective , Crossover, Open-label Study.
Brief Title: A New Application of Amiloride in the Treatment of Patient With Chronic Kidney Disease In Reducing Urinary PROtein
Acronym: ANTI-UPRO
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Guangdong Provincial People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: GGH2016422H
Record Dates: First submitted 2017-05-26; First posted 2017-05-31 (Actual); Last update posted 2020-09-18 (Actual); Status verified 2019-02

CONDITIONS: Chronic Kidney Diseases
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Amiloride; Hydrochlorothiazide

STUDY DESIGN:
Intervention Model Description: All patients need to be on an angiotensin converting enzyme (ACE) inhibitor or an angiotensin receptor blocker (ARB) daily at least four weeks prior to the study. The baseline data would be recorded. Patients enrolled will receive either amiloride or hydrochlorothiazide first for 8 weeks.Then the patients will discontinue amiloride or hydrochlorothiazide for a washout for 4 weeks, but continue with ACEI(angiotensin-converting enzyme inhibitor ) or ARB. After that patients will cross over to receive another medication for another 8 weeks.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- amiloride (Experimental): Amiloride first for 8 weeks, then for a washout for 4 weeks, and cross over to receive hydrochlorothiazide for another 8 weeks
  Interventions: Drug: Amiloride
- hydrochlorothiazide (Active Comparator): hydrochlorothiazide first for 8 weeks, then for a washout for 4 weeks, and cross over to receive amiloride for another 8 weeks.
  Interventions: Drug: Hydrochlorothiazide

INTERVENTIONS:
Drug: Amiloride — Amiloride first for 8 weeks, then for a washout for 4 weeks, and cross over to receive hydrochlorothiazide for another 8 weeks.
  Arms: amiloride
Drug: Hydrochlorothiazide — hydrochlorothiazide first for 8 weeks, then for a washout for 4 weeks, and cross over to receive amiloride for another 8 weeks.
  Arms: hydrochlorothiazide

SUMMARY:
Nowadays, the prevalence of chronic kidney disease (CKD) in China is about 10.8%,and nearly 120 million people suffer from CKD, which has become a serious public health problem in China. Study confirmed that proteinuria is an independent risk factor for the continuous deterioration of glomerular filtration rate (GFR) in patients with CKD. So it is of great significance to explore the strategy of reducing proteinuria.

According to our previous study, Amiloride can inhibit the expression of uPAR in podocytes and reduce proteinuria, This clinical trial aims to evaluate the effect and safety of Amiloride in decreasing proteinuria for patients with Chronic Kidney Disease.

DETAILED DESCRIPTION:
Amiloride is a Na+ channel blocker and has been used as a diuretic. It mainly inhibits the exchange of Na+-K+ and Na+-H+ in the distal tubule and collecting duct of the kidney, thus increasing the excretion of Na+ and water, reducing the excretion of K+ and H+. Recent studies have found a significant increase in urine uPA in patients with massive proteinuria.Urine uPA concentration were positively correlated with urinary protein and decreased with remission of proteinuria. In children and adults with nephrotic syndrome,as well as rat with proteinuria induced by puromycin amino-nucleoside, amiloride can inhibit uPA concentration in urine, which may be one of the mechanisms of amiloride in reducing proteinuria.

This study is a prospective , crossover, open-Label study. All patients need to be on an angiotensin converting enzyme (ACE) inhibitor or an angiotensin receptor blocker (ARB) daily at least four weeks prior to the study. The baseline data would be recorded. Patients enrolled will receive either amiloride or hydrochlorothiazide first for 8 weeks.Hydrochlorothiazide, a similar diuretic as amiloride, but not inhibiting urokinase plasminogen activator receptor (uPAR), will be used as a control. Then the patients will discontinue amiloride or hydrochlorothiazide for a washout for 4 weeks, but continue with the ACE inhibitor or ARB. After that patients will cross over to receive another medication for another 8 weeks. We aim to evaluate the effect and safety of Amiloride in decreasing proteinuria for patients with chronic kidney disease.

ELIGIBILITY:
Inclusion Criteria:

* Patients at the age of more than 14 years old with chronic kidney disease
* Good compliance of treatment
* PCR≥500mg/g.cr ，more than double confirmed
* Patients who written informed consent

Exclusion Criteria:

* less than 14 years of age
* eGFR≤30ml/min.1.73m2；
* poor compliance of treatment
* Previously intolerant or allergic to hydrochlorothiazide
* Patients with history of gout within six months
* Patients with active infection
* Patients with severe cardiopulmonary disease and dysfunction of central nervous system
* history of malignancy
* life expectancy is less than 1 years
* women who are pregnant,lactating and lack of contraception.
* enrolled in other clinical trials within 3 months
* patients who have used immunosuppressive agents or corticosteroids recently or in the past 12 weeks.
* patients without informed consent written or who enable or unwilling to comply with protocol approved by researchers.

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2020-08-01 (Actual); Study Completion 2020-08-01 (Actual)

PRIMARY OUTCOMES:
The remission of proteinuria | after treatment for 12 weeks

SECONDARY OUTCOMES:
estimated Glomerular Filtration Rate | after treatment for 12 weeks
  time to a 50% reduction in baseline estimated Glomerular filtration rate (according to CKD-EPI) and to doubling of baseline creatinine
creatinine | after treatment for 12 weeks
  time to doubling of baseline creatinine
hyperkalemia | at 12 weeks after treatment
  The ratio of hyperkalemia occurred at 12 weeks after treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Nephrology Dept,Guangdong General Hospital, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No